CLINICAL TRIAL: NCT02791958
Title: Pharmacodynamic Equivalence Study of Ramipril 10 mg and Atorvastatin 40 mg Administered as a Cardiovascular Fixed Dose Combination Pill AAR as Compared to Monotherapy With the Reference Products Altace® 10 mg and Lipitor® 40 mg
Brief Title: Pharmacodynamic Equivalence of Ramipril 10 mg and Atorvastatin 40 mg Administered as a Cardiovascular (CV) Polypill Acetylsalicylic Acid-Atorvastatin-Ramipril (AAR) as Compared to Monotherapy
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Ferrer Internacional S.A. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: FCD-PP-1501
Record Dates: First submitted 2016-02-15; First posted 2016-06-07 (Estimated); Last update posted 2017-04-10 (Actual); Status verified 2017-04

CONDITIONS: Hypertension
MeSH Terms: conditions — Hypertension | interventions — Blood Circulation; Atorvastatin; Ramipril

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- CV Fixed Dose Combination Pill AAR (Experimental): Cardiovascular Fixed Dose Combination Pill AAR (acetylsalicylic acid 100 mg, atorvastatin 40 mg and ramipril 10 mg).
  Interventions: Drug: Cardiovascular Fixed Dose Combination Pill AAR
- Atorvastatin (Active Comparator): Atorvastatin 40 mg (Lipitor®).
  Interventions: Drug: Atorvastatin 40 mg
- Ramipril (Active Comparator): Ramipril 10 mg (Altace®).
  Interventions: Drug: Ramipril 10 mg

INTERVENTIONS:
Drug: Cardiovascular Fixed Dose Combination Pill AAR — A once daily oral dose of the Cardiovascular Fixed Dose Combination Pill AAR (acetylsalicylic acid 100 mg, atorvastatin 40 mg and ramipril 10 mg) for 4 weeks.
  Arms: CV Fixed Dose Combination Pill AAR
Drug: Atorvastatin 40 mg — A once daily oral dose of atorvastatin 40 mg (Lipitor®) for 4 weeks
  Arms: Atorvastatin
Drug: Ramipril 10 mg — A once daily oral dose of ramipril 10 mg (Altace®) for 4 weeks
  Arms: Ramipril

SUMMARY:
This study is to compare the pharmacodynamics of a Fixed Dose Combination Pill AAR (acetylsalicylic acid 100 mg, atorvastatin 40 mg and ramipril 10 mg) and the respective reference products, atorvastatin (Lipitor®) 40 mg and ramipril (Altace®) 10 mg.

ELIGIBILITY:
Inclusion Criteria:

* Male or female patients aged ≥18 and <75 years.
* Patients with Stage 1 (SBP/DBP: 140-159/90-99 mmHg) or Stage 2 (SBP/DBP: ≥160/≥100 mmHg) hypertension, either untreated or after a wash out period.
* Patients with an LDL cholesterol level of ≥100 mg/dL and, either untreated or after the wash out period.
* Patients untreated with BP lowering and / or lipid lowering medication
* Patients treated with BP lowering and / or lipid lowering medication can be included if the medication can be safely withdrawn as per physician's judgment.
* Provide written informed consent.

Exclusion Criteria:

* Patients with a BMI of > 35
* SBP < 140 mmHg and DBP < 90 mmHg
* Severe hypertension defined as SBP > 180 mmHg and Diastolic Blood Pressure (DBP) > 110 mmHg
* LDL cholesterol level of <100 mg/dL, either untreated or after the wash out period.
* Serum triglyceride concentration ≥400 mg/dL, either untreated or after the wash out period.
* Patients with a medical condition requiring the chronic pharmacological treatments listed below:

  * Cytochrome P450 3A4 (CYP3A4) inhibitors (eg itraconazole, ketoconazole, erythromycin, clarithromycin, telithromycin, HIV protease inhibitors, and nefazodone).
  * Non-steroidal anti-inflammatory drugs (NSAIDs).
  * K-sparing diuretics.
  * Lithium.
  * Amiodarone and verapamil.
  * Oral anticoagulants (eg, warfarin).
  * Steroids.
  * Digoxin.
  * Gemfibrozil.
  * Niacin.
  * Potassium supplements.
  * Cyclosporine.
  * Danazol.
  * Rifampicin.
* Evidence of any known clinically significant chronic disease
* Patients with renal impairment with Creatinine Clearance (CrCl) < 40 mL/ min/ 1.73 m2
* Creatine phosphokinase (CPK) ≥5 x the upper limit of normal (ULN).
* Alanine aminotransferase (ALT) or aspartate aminotransferase (AST) ≥ 3 x ULN.
* Total bilirubin ≥1.5 x ULN
* Medical history or evidence of drug or alcohol abuse.
* Medical history of gastrointestinal bleeding or gastroduodenal ulcer.
* Presence of secondary dyslipidemia.
* For patients on antihypertensive and/ or cholesterol lowering medication impossibility to withdraw it safely as per physician's judgment
* Previous coronary artery bypass graft (CABG).
* Previous percutaneous transluminal coronary angioplasty (PTCA) with a drug-eluting stent.
* Presence of severe congestive heart failure (New York Heart Classification (NYHC) III IV).
* Prior history of stroke, Transient Ischemic Attack (TIA), Myocardial Infarction (MI), and cardiomyopathy with systolic dysfunction (prior documented Left Ventricular Ejection Fraction (LVEF) < 40%)
* Aspirin induced asthma
* Previous intolerance and/or hypersensitivity to ACE inhibitors, statins and/or salicylates.
* Presence of unstable angina.
* Lab values other than specified out of the central laboratory normal range considered clinically significant.
* Patients and their partners not using effective contraception methods (i.e. intra uterine device (IUD) and condom or diaphragm with spermicide and condom) during the study and for at least one month thereafter, oral contraceptives are allowed.
* Pregnant, lactating, breastfeeding, or intends to become pregnant during the course of the study (females only). All women must have a negative urine pregnancy test at the Screening Visit, be surgically sterile (bilateral tubal ligation, bilateral oophorectomy, or hysterectomy) or have a postmenopausal status (no menses) for at least one year.
* Presence of mental illness limiting the capacity for self-care.
* Presence of major systemic illnesses: renal disease, liver disease, neurological or psychiatric disease.
* Participation, in the 30 days preceding enrolment into the study, in any other clinical study in which investigational or marketed drugs were employed.
* Any other medical condition that in the investigators opinion may interfere with the study procedures and/or evaluations.

Ages: 18 Years to 74 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 528 (Estimated)
Dates: Start 2016-03; Primary Completion 2017-10 (Estimated); Study Completion 2017-10 (Estimated)

PRIMARY OUTCOMES:
Difference in the adjusted mean 24-h systolic blood pressure results using ABPM between the baseline (week 0) and the final visit (week 8). | Measures at baseline visit (week 0) and final visit (week 8).
Difference in LDL cholesterol levels between the baseline (week 4) and the final visit (week 8). | Measures at baseline visit (week 4) and final visit (week 8).

SECONDARY OUTCOMES:
Difference in the adjusted mean 24-h diastolic blood pressure results (using ABPM) between the basal and the final visits. | Measures at baseline visit (week 0) and final visit (week 8).
Difference in the adjusted mean 24-h mean arterial pressure results (using ABPM) between the basal and the final visits. | Measures at baseline visit (week 0) and final visit (week 8).
Difference in the adjusted mean 24-h heart rate results (using ABPM) between the basal and the final visits. | Measures at baseline visit (week 0) and final visit (week 8).
Difference in Very Low-Density Lipoprotein (VLDL) cholesterol levels between the basal and the final visits. | Measures at baseline visit (week 0) and final visit (week 8).
Difference in HDL cholesterol levels between the basal and the final visits. | Measures at baseline visit (week 0) and final visit (week 8).
Difference in total cholesterol levels between the basal and the final visits. | Measures at baseline visit (week 0) and final visit (week 8).
Difference in triglyceride levels between the basal and the final visits. | Measures at baseline visit (week 0) and final visit (week 8).
Incidence of Treatment-Emergent Adverse Events [Safety and Tolerability] | Through study completion, an average of 3 months.
  AEs, clinical laboratory parameters (hematology, clinical chemistry, and urinalysis), vital signs, electrocardiogram (ECG), and physical examination.
  The total number of patients with at least one AE and the number of AEs will be included in listings and tabulations. AEs will be coded using MedDRA, classified by system organ class (SOC) and preferred term and tabulated by intensity and causal relationship for each treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Ronald Surowitz, Principal Investigator — Health Awareness, Inc
Locations (36):
- United States (36):
  - Central Alabama Research, Birmingham, Alabama
  - National Research Institute, Los Angeles, California
  - Clinical Trials Research, Sacramento, California
  - Clinical Trials Investigators, Inc, Tustin, California
  - Infoshpere Clinical Research, Inc, West Hills, California
  - Meridien Research, Bradenton, Florida
  - PAB Clinical Research, Brandon, Florida
  - Clinical Research of South Florida, Coral Gables, Florida
  - Clinical Therapeutics Corporation, Coral Gables, Florida
  - Moonshine Research Center, Inc, Doral, Florida
  - Riverside Clinical Research, Edgewater, Florida
  - Nova Clinical Research Center inc, Hialeah, Florida
  - Dr. John C. Gutleber Weight Loss, Beauty, and Family Practice, Homestead, Florida
  - Westside Center for Clinical Research, Jacksonville, Florida
  - Jacksonville Center for Clinical Research, Jacksonville, Florida
  - Health Awareness, Inc., Jupitor, Florida
  - The Chappel Group Research, Kissimmee, Florida
  - Sunrise Medical Center, Lauderdale Lakes, Florida
  - Progressive Medical Research, Port Orange, Florida
  - Meridien Research, St. Petersburg, Florida
  - Cedar Crosse Research Center, Chicago, Illinois
  - Louisville Metabolic and Atherosclerosis Research, Louisville, Kentucky
  - Clinical Trials of America LA, LLC, Monroe, Louisiana
  - DelRicht Research, New Orleans, Louisiana
  - Bay State Clinical Trials, Inc, Watertown, Massachusetts
  - Clinical Research Source, Perrysburg, Ohio
  - Einstein Clinical Research, Lancaster, South Carolina
  - Punzi Medical Center, Carrollton, Texas
  - Cullen Research, LLC, Houston, Texas
  - Research Trials Worldwide LLC, Humble, Texas
  - Central Texas Health Research, New Braunfels, Texas
  - Deleon Research, PLLC, Plano, Texas
  - Physician PrimeCare Research Institute, PLLC dba H, San Antonio, Texas
  - Diagnostics Research Group, San Antonio, Texas
  - Sylvana Research, San Antonio, Texas
  - Chysalis Clinical Research, St. George, Utah

IPD SHARING:
Plan to Share IPD: No